CLINICAL TRIAL: NCT01775371
Title: Effectiveness and Feasibility of Patient Controlled Analgesia in the ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Jacobi Medical Center (Other); Montefiore Medical Center (Other); University of Pennsylvania (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-485; R01NR013980 (NIH)
Record Dates: First submitted 2012-10-03; First posted 2013-01-25 (Estimated); Results first posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Pain
Keywords: Pain; Emergency; Analgesia; ED patients; acute pain; IV opioid
MeSH Terms: conditions — Pain; Emergencies; Agnosia; Acute Pain | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient Controlled Analgesia (Experimental): PCA (loading dose 0.1 mg/kg morphine and demand dose of 1 mg morphine available every 6 minutes)
  Interventions: Device: Patient controlled analgesia (PCA)
- Usual Care (Active Comparator): Usual opioid analgesia determined by the provider
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Patient controlled analgesia (PCA) — Loading dose 0.1 mg/kg morphine and demand dose of 1 mg morphine available every 6 minutes
  Arms: Patient Controlled Analgesia
Other: Usual Care — Usual opioid analgesia determined by the provider
  Arms: Usual Care

SUMMARY:
Background: Inadequate pain management is common in the Emergency Department (ED). Optimal treatment of pain necessitates titration to effective dose due to the large inter-individual variability in opioid requirement. However nurse administered titration is difficult to provide in this setting due to high patient to nurse and physician ratios and multiple urgent competing patient demands. Patient controlled analgesia (PCA) lets ED patients actively participate in pain management by allowing self-titration to their desired level of pain relief. A tightly controlled randomized clinical trial (RCT) funded by the National Institute of Nursing Research (NINR) recently completed by the investigators group provides promising preliminary support for the efficacy and safety of PCA for patients with abdominal pain at a single ED with a dedicated research nurse and standard loading dose given to all patients. Objective: The overall objective is to provide optimal pain management in the ED. Specific aims: 1)To compare the effectiveness and safety of PCA and non-PCA opioid analgesia when nurses involved in clinical care deliver the intervention to a broad group of ED patients with acute pain at multiple clinical centers. The primary hypothesis is that there will be a greater decline in pain over time and similar safety in patients randomized to receive PCA compared to patients receiving standard opioid analgesia. 2) To describe the feasibility of PCA in terms of patient and provider acceptance, resource utilization and cost associated with PCA. Innovation: PCA represents a novel shift from the current provider-driven model of ED pain management to one in which the patient is an active participant. Few prior studies have evaluated ED PCA and no systematic evaluation of time and resources exists. Methodology: An RCT will be performed at 3 clinical centers. 750 patients with acute pain warranting IV opioid administration will be randomized to receive usual opioid analgesia determined by the provider or PCA (loading dose 0.1 mg/kg morphine and demand dose of 1 mg morphine available every 6 minutes). Pain intensity will be measured by a numerical rating scale (NRS) recorded every half hour up to 2 hours after initial opioid administration. Primary endpoints are rate of change in pain intensity from 30 minutes after initial administration of opioid to 2 hours as suggested by the results of the preliminary study and incidence of adverse events. PCA will also be compared to non-PCA opioid analgesia assessed at the end of the 2 hour study period by patient satisfaction with pain management; registered nurse (RN) assessment of time efficiency/ease of use and satisfaction with pain management; and physician satisfaction with pain management. Resource utilization and cost associated with implementation and use of PCA in the ED setting will be assessed by total Registered nurse (RN) time spent on pain management per patient; pharmacy preparation time per patient; material cost per patient and Registered Nurse and Physician training time necessary for PCA implementation. Significance: If PCA is demonstrated to be effective, safe, and associated with patient and provider acceptance and acceptable resource utilization, it has the potential to significantly improve ED pain management.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65
2. Patient deemed by the ED attending physician to require IV opioid analgesia for pain and for whom the ED Attending Physician would consider using PCA

Exclusion Criteria:

1. Patients requiring initial resuscitation that would preclude the use of PCA
2. Long-term use of prescription or non-prescription opioids now or within the past year
3. Recent opioid use within the past 24 hours
4. Chronic pain syndromes
5. Clinician suspicion of current or past opioid dependence/abuse
6. Altered mental status/Clinical suspicion of intoxication
7. Patients expected to require conscious sedation while in the ED
8. Pregnancy or breast-feeding
9. History of chronic obstructive pulmonary disease, history of sleep apnea syndrome, baseline oxygen saturation (room air) < 97%
10. Systolic blood pressure < 100 mm Hg
11. Use of sedative medications e.g. benzodiazepines, monoamine oxidase inhibitors, phenothiazines, or tricyclic antidepressants.
12. History of renal insufficiency/renal failure
13. Prior allergic reaction to morphine
14. Inability to provide informed consent or inability to understand or operate PCA device
15. Previous entry of patient into study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 636 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Polly Bijur, PhD, Principal Investigator — Albert Einstein College of Medicine; Adrienne Birnbaum, MD, Principal Investigator — Jacobi Medical Center
Locations (3):
- United States (3):
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center - Moses Division, The Bronx, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from April 30, 2013 through February 25, 2016 in the Emergency Departments of three medical centers.
Period: Overall Study
Arm/Group | Patient Controlled Analgesia | Usual Care
Started | 306 | 330
Completed | 306 | 330
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Controlled Analgesia | Usual Care | Total
Number analyzed (Participants) | 306 | 330 | 636
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 306 | 330 | 636
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180 | 202 | 382
  Male | 126 | 128 | 254
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 179 | 205 | 384
  African-American | 69 | 80 | 149
  White | 22 | 25 | 47
  Other | 36 | 20 | 56
Region of Enrollment [Number; unit: participants]
  United States | 306 | 330 | 636
Location of pain [Count of Participants; unit: Participants]
  Abdomen | 239 | 254 | 493
  Other | 67 | 76 | 143
Initial Numerical Rating Scale (NRS) of pain intensity score [Count of Participants; unit: Participants] — A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale. The scale ranged from 0-10 where 0 is no pain and 10 is the worst pain imaginable. Higher numbers on the scale indicate higher pain
  Participants
    NRS Score 3-6 | 6 | 19 | 25
    NRS Score 7 | 29 | 27 | 56
    NRS Score 8 | 47 | 59 | 106
    NRS Score 9 | 57 | 56 | 113
    NRS Score 10 | 167 | 169 | 336
Received non-opioid analgesics before arrival to Emergency Department [Count of Participants; unit: Participants]
  Yes | 86 | 105 | 191
  No | 220 | 225 | 445

OUTCOME MEASURES:

1. Primary Outcome: Rate of Change in Pain Intensity Per Hour
Description: Rate of Change in Numerical Rating Scale (NRS) of Pain per hour where 0 indicates "no pain", 10 indicates "worst possible pain" between 30 minutes and 120 minutes post-baseline i.e. NRS at 30 minutes minus NRS at 120 minutes post-baseline.
Time Frame: 1.5 hours
Population: All patients enrolled
Measure: Mean (95% Confidence Interval); unit: Score on a scale per hour
Arm/Group | Patient Controlled Analgesia | Usual Care
Number analyzed (Participants) | 306 | 330
Score on a scale per hour | 1.3 [1.0 to 1.6] | 0.3 [0.0 to 0.6]
Statistical Analysis 1: Comparison: Patient Controlled Analgesia vs Usual Care; The rate of change of NRS pain scores per hour was calculated using a mixed effects linear model. Time is represented as a linear spline with knot at 30 minutes to support the separate estimation of early and late phase rates of change. Fixed effects in the analysis includes study-group indicator, early and late phase time, and interactions between study-group and time. The principal hypothesis test was a z-test of the coefficient of the study group late phase interaction term; Test type: Superiority; p < 0.001, Z-test 2-sided — The a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [0.6 to 1.5] — The direction of the comparison is the Patient Controlled Analgesia minus the standard care group

2. Secondary Outcome: Number of Participants With One or More Adverse Events
Description: Number of participants with one or more adverse events defined by: oxygen saturation measured by pulse oximetry < 92% for one minute or more, respiratory rate <10 breaths/min counted for 60 seconds, or systolic blood pressure < 90 mm Hg.
Time Frame: 2 hours
Population: All patients
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Controlled Analgesia | Usual Care
Number analyzed (Participants) | 306 | 330
Participants
  One or more adverse events | 7 | 1
  No adverse events | 299 | 329
Statistical Analysis 1: Comparison: Patient Controlled Analgesia vs Usual Care; Test type: Superiority; p = 0.025, Chi-squared

3. Secondary Outcome: Patient Satisfaction With Pain Management
Description: Self report of satisfaction with treatment at120 minutes after baseline
Time Frame: 2 hours
Population: Patients with data at 120 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Controlled Analgesia | Usual Care
Number analyzed (Participants) | 281 | 323
Participants
  Satisfied | 247 | 254
  Dissatisfied or neutral | 34 | 69
Statistical Analysis 1: Comparison: Patient Controlled Analgesia vs Usual Care; Test type: Superiority; p = 0.003, Chi-squared

4. Other Pre Specified Outcome: Nurse Preference for PCA or Conventional Administration of IV Opioids
Description: Single question about preference for PCA versus preference for conventional administration of IV opioids.
Time Frame: 2 hours
Population: All Registered Nurses
Measure: Count of Participants; unit: Participants
Groups:
- All Registered Nurses: All Registered Nurses who treated one or more patients in the study
Arm/Group | All Registered Nurses
Number analyzed (Participants) | 198
Participants
  Prefer Usual Care | 102
  No preference | 56
  Prefer PCA | 40
Statistical Analysis 1: Comparison: All Registered Nurses; These outcomes are based on the nurses who took care of patients in the study; Test type: Other — Responses occur with equal probability; p < 0.001, Chi-squared; One-sample chi-squared test of hypothesis that the responses occur with equal probability

5. Other Pre Specified Outcome: Physician Preference for PCA or Usual Care
Description: Single question about physician preference for PCA or conventional administration of IV opioids
Time Frame: 2 hours
Population: All Physicians who entered one or more patients in each arm of the study
Measure: Count of Participants; unit: Participants
Groups:
- All Physicians: All Physicians who entered one or more patients in each arm of the study
Arm/Group | All Physicians
Number analyzed (Participants) | 143
Participants
  Prefer Usual Care | 25
  No Preference | 49
  Prefer PCA | 69
Statistical Analysis 1: Comparison: All Physicians; This outcome is based on the physicians who took care of the patients in the study; Test type: Other — All responses occur with equal probability; p < 0.001, Chi-squared; One-sample chi-squared test of hypothesis that the responses occur with equal probability

ADVERSE EVENTS:
Time Frame: 2 hours
Description: Need for oxygen supplementation or ventilatory assistance Hypotension requiring fluid administration or vasopressors Administration of naloxone (an opioid reversal agent) Oxygen saturation measured by pulse oximetry < 92% for one minute or more Respiratory rate <10 breaths/min counted for 60 seconds Systolic blood pressure < 90 mm Hg.
Arm/Group | Patient Controlled Analgesia | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/306 | 0/331
Serious Adverse Events (participants affected / at risk) | 0/306 | 0/330
Other Adverse Events (participants affected / at risk) | 7/306 | 1/330
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patient Controlled Analgesia (N=306) | Usual Care (N=330)
Hypotension (Cardiac disorders) | 4 | 0 — Systolic blood pressure < 90 mm Hg.
Oxygen desaturation (Respiratory, thoracic and mediastinal disorders) | 3 | 1 — Oxygen saturation <92%

LIMITATIONS AND CAVEATS:
The full benefit of PCA may accrue over a longer period of time than observed during two-hours. Two-hours not be long enough to capture the full benefit of access to re-dosing in response to the diminishing effect of initial analgesic dose over time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No